CLINICAL TRIAL: NCT00778024
Title: The Objective of This Randomized, Single-dose, Two-way Evaluation is to Compare the Bioequivalence of a Test Fluoxetine HCL Formulation (Ranbaxy Laboratories Limited, Lot No. 6320101) to an Equivalent Oral Dose of the Commercially Available Fluoxetine HCL (Prozac®, Dista Products Company, Lot No 6RK57M) in a Test Population of 36 Adult Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Fluoxetine HCL 40 mg Capsules Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 03197
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: Bioequivalence fluoxetine HCL 40 mg capsules fasting conditions
MeSH Terms: interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): fluoxetine HCL 40 mg capsules of ranbaxy
  Interventions: Drug: fluoxetine HCL 40 mg capsules
- 2 (Active Comparator): PROZAC® 40 mg capsules
  Interventions: Drug: fluoxetine HCL 40 mg capsules

INTERVENTIONS:
Drug: fluoxetine HCL 40 mg capsules

SUMMARY:
The objective of this study is to compare the relative bioavailability of fluoxetine HCL 40 mg capsules (by Ranbaxy Laboratories Limited) with that of PROZAC® 40 mg capsules (by Dista Products Company) following a single oral dose (1 x 40 mg capsule) in healthy, adult subjects under fasting conditions

DETAILED DESCRIPTION:
This is a single-dose, open-label, randomized two-way crossover study to evaluate the bioequivalence of a test formulation, versus an equivalent dose of a commercially available reference drug product, in 36 adult subjects, under fasted conditions. Drug administrations are separated by at least 49 days.

Vital signs (sitting blood pressure and pulse rate) were obtained at baseline (Hour 0), and at post-dose Hours 3, 8, 12, 24, 48, 72, 360, and 1056.

Of the 36 subjects enrolled into the study, 31 subjects completed the study in its entirety. Five (5) subjects were dropped out from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: Male and Female; similar proportion of each preferred.
2. Age: At least 18 years.
3. Qualifying subjects must be in good health and physical condition as determined by medical history, complete physical examination, and laboratory tests, all obtained within four (4) weeks prior to study start. The subject may not have a history of significant past illness expected to affect the investigation. The normal status of subjects will be confirmed by the following procedures:

   • Laboratory Tests: Hemoglobin, hematocrit, RBC, WBC, differential count, serum electrolytes (Na, K, CL), fasting blood glucose, BUN, bilirubin, creatinine, AST, ALT, LD, alkaline phosphatase, and urinalysis. HIV, Hepatitis B, Hepatitis C, and drugs of abuse testing will be done for screening purposes only. Urine drugs of abuse testing will be repeated at each check-in. Female subjects will have a serum pregnancy test done at screening and urine pregnancy test prior to each study period at check-in. Laboratory values which are greater than :E20% of the normal range will not qualify unless specifically accepted (with comment) by the Principal Investigator. Results of HIV, Hepatitis B, Hepatitis C, and drugs of abuse must be negative or non-reactive for the subject to qualify for the study.

   • Electrocardiogram: A 12-lead electrocardiogram (ECG) will be obtained for all subjects. The original tracings, plus interpretation, will be included in the case report form packet.
4. Subjects must read and sign the Consent Form.

Exclusion Criteria:

1. Subjects not complying with the above inclusion criteria must be excluded from the study.
2. In addition, any one of the conditions listed below will exclude a subject from the study:

   * History of treatment for alcoholism, substance abuse, or drug abuse within past 24 months.
   * History of malignancy, stroke, diabetes, cardiac, renal or liver disease, or other serious illness.
   * History of GERD (gastroesophageal reflux disease), malabsorption syndrome, colon cancer, or chronic colitis, including Crohn's disease.
   * History of treatment for astlzurta within the past five (5) years.
   * History of neurological impairment.
   * History of seizures.
   * History of Parkinson's Disease.
   * History of diabetes mellitus.
   * Females who are pregnant or lactating.
   * History of hypersensitivity to fluoxetine HCL, or any serotonin reuptake inhibitor.
3. Conditions upon screening which might contraindicate or require that caution be used in the administration of fluoxetlne HCL, including:

   * Sitting systolic blood pressure below 90 mm Hg, or diastolic Pressure below 50 mm Hg.
   * Heart rate less than 50 beats per minute after a 5-minute rest
4. Inability to read and/or sign the consent form.
5. Treatment with any other investigational drug during the four (4) weeks prior to the initial dosing for this study.
6. Subjects who have donated blood within four (4) weeks prior to the Initial dosing for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2003-08; Primary Completion 2003-10 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Gateway medical research, Saint Charles, Missouri, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html